CLINICAL TRIAL: NCT05662137
Title: The Effect of Recognition and Expression of Emotions Program Applied to Schizophrenia Patients Applying to Community Mental Health Center on Alexithymia and Emotion Expression
Brief Title: The Effect of Recognition and Expression of Emotions Program Applied to Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: sınopUadeviye-1
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia; Alexithymia; Emotion, Expressed
Keywords: Alexithymia; Schizophrenia; Emotion, Expressed
MeSH Terms: conditions — Schizophrenia; Affective Symptoms | interventions — Gene Expression

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): At the beginning of the study, data collection tools Personal Information Form, Expression of Emotions Scale, Toronto Alexithymia Scale, Positive and Negative Syndrome Scale will be applied to the control group.
  No intervention will be made in the control group. Measurement tools will be applied for the posttest. Emotional Expression Scale, Toronto Alexithymia Scale and Positive and Negative Syndrome Scale will be reapplied 1 month after the last session.
- Experimental group (Experimental): Emotion recognition and expression program is aimed to be carried out in 8-week sessions for schizophrenia patients included in the experimental group. Personal Information Form, Expression of Emotions Scale, Toronto Alexithymia Scale, Positive and Negative Syndrome Scale will be applied to the experiment. The principal investigator will lead the structured group sessions as the group leader.
  The principal investigator will lead the structured group sessions as the group leader.
  Each group is planned to be 60-90 minutes. Before sessions, participants are taken from their previous session's emotions so far. Homework is discussed by providing recall of the topic from the previous session, and then the current topic is moved on. At the end of each session, a general summary and evaluation is made. After the sessions in the research, measurement tools will be applied for the posttest. It will be reapplied 1 month after the last session.
  Interventions: Behavioral: Emotions Recognition and Expression

INTERVENTIONS:
Behavioral: Emotions Recognition and Expression — Emotion recognition and expression program consisting of 8 sessions will be used. In this program, patients will have the opportunity to describe their emotions, explain emotions that are difficult to express such as anger, sadness, shame, guilt, and discuss the consequences of suppressed emotions.
  Arms: Experimental group

SUMMARY:
As a result of the positive and negative symptoms that occur in schizophrenia, patients with schizophrenia may experience negative emotions more frequently than individuals with other mental problems. Since these emotions can trigger psychotic symptoms, there is a need to develop effective emotion regulation strategies to be applied to patients with schizophrenia.

Aim: In this study, it was aimed to examine the effect of emotion recognition and expression program on alexithymia and emotion expression in patients with schizophrenia.

DETAILED DESCRIPTION:
Method: Fifty schizophrenic patients who regularly receive outpatient treatment at Sinop Community Mental Health Center will form the universe of the study. Individuals over the age of 18 who have schizophrenia, do not have mental retardation, have no comprehension and hearing problems, have insight, and are in remission will be included in the study. Individuals who meet the study criteria will be divided into experimental and control groups as 22 experimental and 22 control groups. The emotion recognition and expression program prepared by the researchers in line with the literature will be applied to the experimental group for 8 weeks. Personal Information Form, Expression of Emotions Scale, Positive and Negative Syndrome Scale and Toronto Alexithymia Scale were planned to be applied to the experimental and control groups in the pre-test, post-test and follow-up. Follow-up will take place one month after the last session of the study. Psychosocial interventions applied to patients with schizophrenia help patients to increase their level of well-being and quality of life, to decrease negative and positive symptoms by increasing social functionality, to participate in social life, to be an autonomous individual and to prevent stigma. In line with psychosocial interventions, it is thought that the this program to be applied to the patients in this study will basically contribute to the individual patients' ability to recognize their emotions, discuss their emotions, regulate their emotion intensities, and express their emotions. Due to the impact that this program will have on the individual, it is believed that it will have positive results not only for schizophrenia patients, but also for the individuals with whom the patients interact, their relatives and even the society.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had received a diagnosis of schizophrenia and comes to the Community Mental Health Center regularly,
* Being able to read and communicate
* Being 18 years of age or older,
* Not having mental retardation,
* Not having insight, understanding, hearing problems,
* Being in remission,
* Volunteering to study

Exclusion Criteria:

* Not diagnosed with clinical schizophrenia,
* Being under the age of 18,
* Having mental retardation,
* Having no insight,
* Not understanding and hearing,
* Not in remission
* Refusing to participate in the study
* Stop studying at any stage of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Emotion Recognition and Expression | One day
  Expression of Emotions Scale is used to measure the state of expression of emotions. The scale was developed by King and Emmons (1990), and its Turkish validity and reliability were verified by Kuzucu (2011). The measurement tool consists of a total of 16 items and 3 sub-dimensions. It has positive, negative and closeness sub-dimensions. It is a 7-point Likert type scale .The scores to be taken from the scale vary between 15 and 105, and as the scores obtained increase, it is seen that the tendency of the individual to express emotion increases. The scale provides information about expressing emotions both in interpersonal relationships and independent of interpersonal relationships. A high score indicates a high tendency to express emotions.
Alexithymia | One day
  Toronto Alexithymia Scale (TAS): The scale was developed by Bagby et al. (1994) Güleç et al. (2009) adapted into Turkish. The scale consists of 20 items, has three sub-dimensions and is in a 5-point Likert type. High scores indicate high alexithymic level. There are sub-dimensions of difficulty in recognizing emotions, difficulty in putting emotions into words, and extroverted thinking.
Positive and Negative Syndrome | One day
  Positive and Negative Syndrome Scale (PANNS): The scale evaluating positive and negative symptoms in schizophrenia was developed by Kay et al (1987) and Kostakoğlu et al. It was adapted into Turkish by (1999). Consisting of 30 items, the scale has three sub-dimensions. A 7-point severity assessment is carried out. Seven of the items of the scale belong to the positive symptoms subscale, seven to the negative symptoms subscale, and the remaining sixteen to the general psychopathology subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Adeviye AYDIN, PhD, Principal Investigator — Sinop University
Locations (1):
- Sinop Community Mental Health Center, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No